CLINICAL TRIAL: NCT06409182
Title: A Prospective Pilot Study to Evaluate the Diagnostic Performance of a Wireless Sensor Capsule in Detection of Upper Gastrointestinal Bleeding
Brief Title: A Prospective Pilot Study to Evaluate the Diagnostic Performance of a Wireless Sensor Capsule in Detection of UGIB
Acronym: HemoPill
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Louis Ho Shing Lau, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023.549
Record Dates: First submitted 2024-02-01; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: UGI Bleed

STUDY DESIGN:
Intervention Model Description: Patient will swallow wireless sensor capsule to determine if there's
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemopill (Experimental): HemoPill® acute capsule (Ovesco Endoscopy, Tuebingen, Germany) is a swallowable, wireless, sensor capsule designed for in vivo detection of liquid blood or hematin. The capsule has integrated optical microsensor for blood detection, by transmitting red and violet light via LEDs. It allows the detection of blood by photometric measuring method, in small volumes or in unprepared digestive tract. The dimensions of the capsules are 7.0mm x 26.3mm. The maximal examination time is 9 hours. The HemoPill® receiver is a portable receiver for displaying and storing measured values from the HemoPill® acute capsule. It allows a real-time, wireless, telemetric data transmission. Once activated, the HemoPill® acute capsule can be swallowed by patients with real-time measurement of HemoPill® Indicator (HI). An HI value in the red range suggests a positive finding - liquid blood or hematin has been detected.
  Interventions: Device: Hemopill

INTERVENTIONS:
Device: Hemopill — HemoPill® acute capsule (Ovesco Endoscopy, Tuebingen, Germany) is a swallowable, wireless, sensor capsule designed for in vivo detection of liquid blood or hematin. The capsule has integrated optical microsensor for blood detection, by transmitting red and violet light via LEDs. It allows the detection of blood by photometric measuring method, in small volumes or in unprepared digestive tract. The dimensions of the capsules are 7.0mm x 26.3mm. The maximal examination time is 9 hours. The HemoPill® receiver is a portable receiver for displaying and storing measured values from the HemoPill® acute capsule. It allows a real-time, wireless, telemetric data transmission. Once activated, the HemoPill® acute capsule can be swallowed by patients with real-time measurement of HemoPill® Indicator (HI). An HI value in the red range suggests a positive finding - liquid blood or hematin has been detected.

SUMMARY:
It is a single-center, prospective study, which will be conducted in a tertiary academic hospital (Prince of Wales Hospital). All subjects will undergo a paired examination of HemoPill® acute capsule and oesophago-gastro-duodenoscopy (OGD).

DETAILED DESCRIPTION:
It is a single-center, prospective study, which will be conducted in a tertiary academic hospital (Prince of Wales Hospital). All subjects will undergo a paired examination of HemoPill® acute capsule and oesophago-gastro-duodenoscopy (OGD).

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible if:

* They have symptoms and signs of suspected UGIB (melena, per rectal bleeding, coffee ground vomiting, history of hematemesis);
* They will undergo OGD within 24 hours;
* Written consent obtained.

Exclusion Criteria:

Subjects will be excluded from the study if they have any of the followings:

* Contraindications for OGD (e.g. respiratory failure, suspected perforation);
* Contraindications for capsule endoscopy (e.g. known gastrointestinal obstruction or stricture, severe dysphagia, impaired consciousness);
* Cardiac pacemaker or implanted electromedical devices;
* History of gastrectomy or bowel resection;
* Active ongoing fresh hematemesis;
* Unstable hemodynamics despite adequate resuscitation;
* Advanced comorbidities (defined as American Society of Anesthesiologists grade 4 or above);
* Pregnancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-11-29 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Area under the ROC curve | duration of study, 2 hours
  The primary endpoint is the area-under-the-ROC curve (AUC) for HemoPill® capsule, which is defined by the true positive and false positive rates of HI signals.

SECONDARY OUTCOMES:
Sensitivity | duration of study, 2 hours
  Sensitivity of Hemopill
Specificity | duration of study, 2 hours
  Specificity of Hemopill
Positive predictive value | duration of study, 2 hours
  Positive predictive value of Hemopill
Negative predictive value | duration of study, 2 hours
  Negative predicitive value of Hemopill
Technical success rate | duration of study, 2 hours
  Technical success rate of Hemopill
Adverse event rate | duration of study, 2 hours
  Adverse event rate of Hemopill
Time to a positive HI signal | duration of study, 2 hours
  Time to a positive HI signal of Hemopill
Time to OGD from Hemopill capsule examination | duration of study, 2 hours
  Time to OGD from Hemopill capsule examination

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No